CLINICAL TRIAL: NCT05409651
Title: Phenotyping Mitochondrial and Immune Dysfunction in POTS With Targeted Clinical Intervention.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Dysautonomia International (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 802200
Record Dates: First submitted 2022-05-16; First posted 2022-06-08 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Time-Restricted Eating; Intermittent fasting; POTS; Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Intermittent Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time restricted eating (Experimental): Everyone in this arm will implement a daily 8-10-hour window within which they must consume their calories. They will also be required to log their caloric intake through the use of a smartphone app.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Participants in this arm will adhere to a daily, consistent 8-10-hr eating window for the course of the study.
  Other Names: TRE

SUMMARY:
The mechanisms underlying POTS are not well understood. Though heterogeneous in nature, patients often present with symptoms that include fatigue, orthostatic lightheadedness and tachycardia, "brain fog", shortness of breath, and sleep disruption. The central mediator that links observations in disease entities similar to POTS is energy use and balance driven by mitochondrial health. Mitochondrial dysfunction (i.e. respiration defects, reactive oxygen species (ROS) generation, and structural abnormalities) are hallmarks of currently defined syndromes that resemble POTS symptomatology. Many patients with POTS have underlying immune system dysfunction, which, when treated, may improve the patient's overall health. Though autoimmunity has been demonstrated in POTS, overall immune dysregulation may be broader and include immune cell exhaustion and persistent inflammatory cytokine responses. Immune dysfunction including cellular exhaustion and persistent inflammation has been linked to mitochondrial function. Therefore, we hypothesize that a unifying feature of POTS results from latent or continued mitochondrial/immune dysfunction which then impacts multi-organ energy imbalance and immune homeostasis. Understanding and targeting mitochondria utilizing established, novel, and directed approaches including time-restricted eating (TRE) will help to unravel common etiologies and help us to better diagnose, manage, and treat POTS.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old
2. POTS, as defined by the presence of any of the following criteria:

   * For patients age 20 or older, increase in heart rate ≥ 30 bpm within ten minutes of upright posture (tilt test or standing) from a supine position (For patients age 18-19, heart rate increase must be >40 bpm)
   * Associated with related symptoms that are worse with upright posture and that improve with recumbency
   * Chronic symptoms that have lasted for longer than six months
   * In the absence of other disorders, medications, or functional states that are known to predispose to orthostatic tachycardia
3. Baseline eating period > 12-hour window

   Exclusion Criteria:
4. Taking insulin within the last 6 months.
5. Manifest diabetes, defined as HbA1c > 7.0% given a 0.3% margin of error in lab readings, or diagnosis of diabetes.
6. Known inflammatory and/or rheumatologic disease.
7. Active tobacco abuse or illicit drug use or history of treatment for alcohol abuse.
8. Pregnant or breast-feeding women.
9. Shift workers with variable (e.g. nocturnal) hours.
10. Caregivers for dependents requiring frequent nocturnal care/sleep interruptions.
11. Planned travel to a time zone with greater than a 3-hour difference during study period.
12. History of a major adverse cardiovascular event within the past 1 year (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA)).
13. Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria).
14. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
15. History of adrenal disease.
16. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
17. Known history of type I diabetes.
18. History of eating disorder.
19. History of cirrhosis.
20. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
21. History of HIV/AIDS.
22. Currently enrolled in a weight-loss or weight-management program.
23. On a special or prescribed diet for other reasons (e.g. Celiac disease).
24. Currently taking any medication that is meant for, or has known effect on, appetite.
25. Any history of surgical intervention for weight management.
26. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).
27. A score of >16 on the Epworth Sleepiness Scale (ESS).
28. Depression determined by the Beck Depression Inventory (BDI-II) (unless previously diagnosed and well-controlled)
29. Failure to use the smartphone app for documentation (defined as <2 meals/day for ≥3 days during baseline).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Conduct a pilot clinical trial with POTS patients to assess if TRE can improve Quality of Life. | Change from Baseline quality of life questionnaire at 14 weeks
  Intervention with TRE will significantly improve quality of life (QOL). We will conduct a 12-week intervention with POTS patients to assess the impact of TRE on QOL (primary endpoint) utilizing the quality of life questionnaire SF-36..

OTHER OUTCOMES:
Exploratory Outcome: Characterize mitochondrial function in POTS patients | Change from Baseline mitochondrial function at 14 weeks
  Mitochondrial damage is a common feature of POTS regardless of triggers, comorbidities, and heterogeneity. We will test this hypothesis by assessing blood-based markers of mitochondrial function in patients with POTS and compare to banked healthy controls.
Exploratory Outcome: Assess whether POTS patients demonstrate persistent inflammatory responses and immune cell exhaustion | Change from Baseline immune response at 14 weeks
  Immune homeostasis is disrupted in POTS leading to aberrant persistent cytokine responses and immune cell (T, B, NK cell) exhaustion. We will test immune exhaustion and persistent inflammation through flow cytometry of peripheral blood cells from patients with POTS as well as perform serum multiplex ELISA of cytokines and compare them with banked controls.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — Professor of Medicine; Taylor Doherty, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States